CLINICAL TRIAL: NCT01976936
Title: A Phase 2 Safety Study in Which Ischemic Stroke Patients Will be Randomized Within 24 Hours of Symptom Onset to Placebo or Oral Lovastatin 640 mg Per Day for 3 Days.
Brief Title: Neuroprotection With Statin Therapy for Acute Recovery Trial Phase 2
Acronym: NeuSTART2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAD9004; 2P50NS049060 (NIH)
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Results first posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Rhabdomyolysis; Jaundice
Keywords: Stroke; Rhabdomyolysis; Jaundice
MeSH Terms: conditions — Stroke; Rhabdomyolysis; Jaundice | interventions — Lovastatin; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High Dose Lovastatin (Experimental): High dose lovastatin (640 mg daily for three days) will be administered orally
  Interventions: Drug: High Dose Lovastatin
- Low Dose Lovastatin (Active Comparator): Lovastatin 80 mg daily for three days will be administered orally to patients who were taking statin therapy at the time of enrolment
  Interventions: Drug: Low Dose Lovastatin
- Placebo (Placebo Comparator): Placebo will be administered orally to patients who were NOT taking statin therapy at the time of enrolment
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Low Dose Lovastatin — 80 mg daily for 3 days
  Other Names: Mevacor
  Arms: Low Dose Lovastatin
Other: Placebo — Placebo for 3 days
  Other Names: microcrystalline cellulose
  Arms: Placebo
Drug: High Dose Lovastatin — 640 mg daily for 3 days
  Other Names: Mevacor
  Arms: High Dose Lovastatin

SUMMARY:
This trial will be a phase 2 randomized safety study in which ischemic stroke patients will be randomly assigned within 24 hours of symptom onset to placebo or standard dose lovastatin versus short-term high-dose lovastatin 640 mg per day for 3 days. The primary outcome of this Phase 2 study will be musculoskeletal and hepatic toxicity, defined by clinical and laboratory criteria, with a 3-month follow-up period (± 1 week). Secondary outcomes will include neurological outcome (National Institute of Health (NIH) Stroke Scale), functional outcomes (Barthel Index), and handicap (modified Rankin scores). Effects on inflammatory markers and lipid levels will also be assessed.

DETAILED DESCRIPTION:
This is a phase 2 randomized, blinded and controlled safety study in patients with ischemic stroke. The time window for enrollment will be within 0-24 hours of symptom onset. For patients who are found with the stroke on awakening, it will be assumed that the stroke occurred the last time that the patient was known to be normal. All patients will be identified by the stroke acute care team in the emergency room of the participating centers, or in some cases, on the floor services of the hospital (i.e., for patients with stroke occurring in hospital). If preliminary data indicate that the patient meets eligibility criteria the patient (or legally authorized representative) will be approached about participation in the study, and consent obtained. Surrogate consent will be allowed at centers at which this is permitted according to regulations. Patients who are consented through a surrogate and subsequently regain capacity, will be approached and reconsented to continue in the study.

The intervention chosen for this trial is either (1) placebo for patients not taking a statin at the time of admission OR lovastatin 80 mg in place of their regular statin for patients taking a statin (atorvastatin, simvastatin, rosuvastatin, pravastatin, fluvastatin, lovastatin) at time of enrolment VERSUS (2) oral lovastatin at dosage of 640 mg daily for 3 days. The time of first dose will be considered time 0. Patients will be administered the total daily dose in four daily divided doses (i.e., QID schedule). After the initial 3 days of acute dosage, all patients will receive statin therapy at the discretion of their treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18
2. Satisfies the criteria for ischemic stroke: acute focal neurological deficit of likely ischemic vascular origin.
3. Patient or legally authorized representative has provided written informed consent prior to study entry. Patient who regains capacity provides his/her written consent to remain in the study.
4. Patient can receive the first treatment dose within 0-24 hours of stroke onset. For patients found with stroke on awakening, it will be assumed that the stroke occurred the last time that the patient was known to be normal.
5. Patient has pretreatment brain CT scan compatible with ischemic stroke and excludes hemorrhagic and non-vascular etiologies of symptoms.
6. Patients taking statins at time of stroke may be included.
7. Patients receiving standard dose intravenous tPA or mechanical interventional procedures may be enrolled.

Exclusion Criteria:

1. Brain imaging study shows a lesion other than ischemic stroke that could explain patient's symptoms (intracranial or subarachnoid hemorrhage, arteriovenous malformation, aneurysm, multiple sclerosis, tumor, abscess or other). Asymptomatic meningiomas are allowed.
2. Mild stroke, defined as NIH Stroke Scale <2.
3. Weight < 50 kg.
4. Patient is comatose, regardless of etiology (> 4 points on the first three items of the NIHSS).
5. History of intolerance or allergic reaction to any statins (myotoxicity, hepatic dysfunction, rash, etc.)
6. Use of drugs within past 30 days that utilize the cytochrome CYP3A pathway (cyclosporine, itraconazole, ketoconazole, erythromycin, clarithromycin, nefazodone, posaconazole, voriconazole, dronedarone, diltiazem, colchicine and ranolazine).
7. Use of drugs within past 30 days that increase risk of myotoxicity with statins (gemfibrozil, other fibrates, niacin, amiodarone, verapamil).
8. Baseline major electrolyte disturbances (sodium <125 or >150, potassium <3.0 or >5.5).
9. Recent major trauma (<3 months).
10. Hypothermia (body temperature < 96F).
11. Baseline hypoxia (defined as oxygen saturation <92% on room air).
12. History of likely or proven systemic viral infection within 30 days.
13. Known HIV infection or use of protease inhibitors.
14. Endocarditis likely as cause of stroke.
15. Mitochondrial disorder likely as cause of stroke.
16. Pregnancy or lactation.
17. History of rhabdomyolysis, myopathy, or other severe muscle disease.
18. History of hepatitis, decompensated liver disease (ascites, bleeding varices or encephalopathy), or liver failure.
19. Liver function tests (ALT, AST) > 2 X upper limit of normal.
20. Unstable cardiovascular (includes uncontrolled hypertension), pulmonary, gastrointestinal, hepatic or musculoskeletal disease.
21. Patient has evidence of severe congestive heart failure or has history of end-stage cardiovascular disease (e.g. CHF NYHA Class III or IV or unstable angina).
22. Abnormal ECG showing: Hemodynamically significant arrhythmia or frequent PVCs (>5/minute) (controlled atrial arrhythmia will not be an exclusion); evidence of acute myocardial infarction; Mobitz Type II 2nd degree AV block or 3rd degree AV block; ventricular tachycardia or ventricular fibrillation.
23. Significant renal insufficiency, indicated by serum creatinine >2.0 mg/dl.
24. Hypoglycemia (glucose < 60 mg/dl) or diabetic ketoacidosis unresponsive to therapy.
25. Any of these hematologic abnormalities: WBC <3.0 x 103/mm3; Platelet count <50,000/mm3
26. Received an investigational drug within 30 days.
27. Severe behavioral or social problems that may interfere with the conduct of clinical study procedures.
28. Patient unlikely, in the investigator's opinion, to complete the study and return for follow-up visits for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Elkind, MD, MS, Principal Investigator — Columbia University
Locations (7):
- United States (7):
  - University of California, Los Angeles Stroke Network, Los Angeles, California
  - Jackson Memorial Hospital, Miami, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Mount Sinai School of Medicine, New York, New York
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard: Includes individuals on placebo or 80mg of Lovastatin
- High Dose: Includes individuals on 640mg of Lovastatin
Period: Overall Study
Arm/Group | Standard | High Dose
Started | 81 | 81
Completed | 72 | 77
Not Completed | 9 | 4
Not completed — Did not receive at least 9 doses | 9 | 4

BASELINE CHARACTERISTICS:
Population: Includes all individuals who received treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard | High Dose | Total
Number analyzed (Participants) | 81 | 81 | 162
Age, Customized [Count of Participants; unit: Participants]
  ≥ 18 years | 81 | 81 | 162
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 36 | 75
  Male | 42 | 45 | 87

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Participants With an Increase in Liver Function Tests (LFTs)
Description: The development of clinical or laboratory evidence of major hepatic toxicity within 7 days of treatment onset or the development of clinical or laboratory evidence of rhabdomyolysis within 7 days of treatment onset.
  The primary safety outcome will be defined as:
  Liver toxicity: LFT increase at any time point > 3X upper limit of normal or development of jaundice, otherwise unexplained coagulopathy, or other clinical evidence of hepatitis or liver failure;
  or
  Muscle toxicity: An increase in CK (Creatine Kinase) at any time point > 10 X upper limit of normal, or clinical evidence of muscle pain or weakness not related to the stroke and associated with CK > 5 X upper limit of normal.
Time Frame: 7 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard | High Dose
Number analyzed (Participants) | 81 | 81
Participants | 1 | 2

2. Secondary Outcome: Mean Score on NIH Stroke Scale (NIHSS)
Description: The National Institutes of Health Stroke Scale (NIHSS) is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke and to measure neurological outcomes. The NIHSS is composed of 11 items, with a score range of 0-42. Higher scores indicate greater impairment caused by a stroke.
Time Frame: 90 days
Population: Only includes individuals who completed the NIHSS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard | High Dose
Number analyzed (Participants) | 57 | 62
score on a scale | 2.5 (3.3) | 3.3 (4.2)

3. Secondary Outcome: Total Number of Participants With a Barthel Index Score > 95
Description: The Barthel Index will be used to measure functional outcomes by counting the total number of individuals with a Barthel index score greater than or equal to 95. Numerical scores based on whether an individual requires physical assistance to perform the task or can complete it independently. An individual scoring 0 points would be dependent in all assessed activities of daily living, whereas a score of 100 would reflect independence in these activities, indicative of a better outcome.
Time Frame: 90 days
Population: Only includes individuals who completed Barthel Index.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard | High Dose
Number analyzed (Participants) | 65 | 70
Participants | 46 | 38

4. Secondary Outcome: Total Number of Participants With a Modified Rankin Score of 0-1
Description: The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It will be used as a measure of handicap by looking at the total number of individuals with a score of 0-1. The scale runs from 0-6, running from perfect health without symptoms (score of 0) to death (score of 6). A score of 0 indicates a better outcome.
Time Frame: 90 days
Population: Only analyzed from individuals with modified rankin scale data at Day 90.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard | High Dose
Number analyzed (Participants) | 67 | 72
Participants | 29 | 31

ADVERSE EVENTS:
Time Frame: Data was collected up to 1 year after data collection for all outcome measures.
Description: Data regarding all non-serious and serious adverse events were collected according to the system type per kit used by subjects, so safety data is reported as a combined summary (incorporates all arms) and not reported per arm. The adverse event data is only available as a summary (arms combined) and cannot be separated by arm as the study has closed with the Institutional Review Board (IRB) and additional analysis cannot be performed.
Groups:
- All Subjects Treated: This includes all individuals who began treatment with the study medication.
Arm/Group | All Subjects Treated
All-Cause Mortality (participants affected / at risk) | 2/162
Serious Adverse Events (participants affected / at risk) | 62/162
Other Adverse Events (participants affected / at risk) | 8/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects Treated (N=162)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 8 (9)
Infections and Infestations (Infections and infestations) | 37 (41)
Cardiac disorders (Cardiac disorders) | 35 (36)
Nervous system disorder (Nervous system disorders) | 48 (54)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 10 (11)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 8 (9)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 3 (3)
Hepatobiliary disorders (Hepatobiliary disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) — This includes cysts and polyps
Gastrointestinal disorders (Gastrointestinal disorders) | 22 (26)
Surgical and medical procedures (Surgical and medical procedures) | 15 (17)
Vascular disorders (Vascular disorders) | 13 (15)
Investigations (Investigations) | 30 (40)
Psychiatric disorders (Psychiatric disorders) | 9 (9)
Renal and urinary disorders (Renal and urinary disorders) | 5 (6)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 2 (2)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 16 (19)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 6 (6)
Immune system disorders (Immune system disorders) | 2 (2)
Eye disorders (Eye disorders) | 1 (1)
General disorders and administration site conditions (General disorders) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects Treated (N=162)
Infections and Infestations (Infections and infestations) | 3 (3)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (2)
Cardiac disorders (Cardiac disorders) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 1 (1)
Nervous system disorders (Nervous system disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Investigations (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes